CLINICAL TRIAL: NCT02386618
Title: Endoscopic Treatment for Local Residual Neoplasia After Endoscopic Mucosal Resection of the Colorectal Lateral Spreading Tumors (LST)
Brief Title: Endoscopic Treatment for Local Residual Neoplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitkovice Hospital (Other)
Responsible Party: Principal Investigator, Premysl Falt, M.D., Ph.D., MUDr. Premysl Falt, Vitkovice Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DDC VN 07
Record Dates: First submitted 2013-09-19; First posted 2015-03-12 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; laterally spreading tumors; endoscopic mucosal resestion; local residual neoplasia
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Local residual neoplasia (Other): Patients with local residual neoplasia in 3 months after endoscopic resection of colorectal lateral spreading tumors diagnosed endoscopically and/or histologically
  Interventions: Procedure: Standardized endoscopic treatment of local residual neoplasia

INTERVENTIONS:
Procedure: Standardized endoscopic treatment of local residual neoplasia — Endoscopic treatment will be performed according to the type of local residual neoplasia (LRN): A - endoscopically negative scar and neoplastic tissue found only in biopsy specimens - treatment by argon plasmacoagulation, B - endoscopically aparent LRN < 5 mm - forceps biopsy + argon plasmacoagulation, C - endoscopically evident LRN > 5 mm + lifting during submucosal injection - endoscopic mucosal resectio + argon plasmacoagulation, D - endoscopically evident LRN > 5 mm + non-lifting during submucosal injection - endoscopic submucosal disection (ESD) or surgical resection

SUMMARY:
Endoscopic mucosal resection (EMR) is considered to be a gold standard of therapy of colorectal lateral spreading tumors (LST) without significant risk for lymphatic spread. According to the investigators previous study, local residual neoplasia (LRN) after conventional endoscopic mucosal resection (EMR)occurs in up to 21% of cases. Endoscopic therapy of LRN was not sufficient in 53 % and has not been standardized yet.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years
* patients with local residual neoplasia in scar in three months after endoscopic mucosal resection for laterally spreading tumor (0-IIa > 10 mm)
* signed informed consent

Exclusion Criteria:

* incomplete endoscopic mucosal resection
* previous therapy for local residual neoplasia
* difficult or impossible localization of post-EMR scar

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Efficacy of endoscopic treatment od local residual neoplasia (absence of neoplastic tissue in post-EMR scar proven by endoscopic and histologic examination) | 6 months
  Efficacious endoscopic treatment is defined as absence of neoplastic tissue in post-EMR scar proven by endoscopic and histologic examination in 6 months after endoscopic treatment od local residual neoplasia.

CONTACTS AND LOCATIONS:
Overall Officials: Premysl Falt, MD, PhD, Principal Investigator — Vitkovice Hospital, Ostrava
Locations (1):
- Vitkovice Hospital, Ostrava, Czechia